CLINICAL TRIAL: NCT05036291
Title: A Phase 1, Open-label, Multicenter Study to Assess the Safety, Tolerability, and Pharmacokinetics of NB004 Administered as Monotherapy or Combination Therapy in Subjects With Advanced Solid Tumors
Brief Title: A Study of NB004 as Monotherapy or Combination Therapy in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ningbo Newbay Technology Development Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB004-01
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NB004 (Experimental): Part1: Dose escalation phase of study drug NB004 monotherapy:
  Part 2: Dose Escalation Phase for the NB004 in combination with Sotorasib:
  Part 3: COMBO Dose Expansion Phase for the NB004 in combination with Sotorasib:
  Interventions: Drug: NB004 tablets

INTERVENTIONS:
Drug: NB004 tablets — Part1: Dose escalation phase of study drug NB004 monotherapy:
  Drug: NB004 tablets
  NB004 tablets will be administered orally once daily for repeated 28-day cycles until discontinuation criteria are met.
  Part 2: Dose Escalation Phase/ COMBO Dose Expansion Phase for the NB004 in combination with Sotorasib:
  Drug: NB004 tablets & Sotorasib
  NB004 tablets will be administered orally once a daily for repeated 21-day cycles until discontinuation criteria are met.
  Sotorasib will be administered with the recommended dosage per prescribing information approved by the FDA
  Part 3: Dose Escalation Phase/ COMBO Dose Expansion Phase for the NB004 in combination with Sotorasib:
  Drug: NB004 tablets & Sotorasib
  NB004 tablets will be administered orally once daily for repeated 21-day cycles until discontinuation criteria are met.
  Sotorasib will be administered with the recommended dosage per prescribing information approved by the FDA .
  Other Names: Sotorasib

SUMMARY:
This is a Phase 1, Open-label, Multicenter Study to Assess the Safety, Tolerability, and Pharmacokinetics of NB004 Administered as Monotherapy or Combination Therapy in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
This study is a Phase 1, open-label, multicenter study of NB004 administered orally in patients with histologically and/or cytologically confirmed diagnosis of advanced solid tumors that are metastatic for which all standard treatment options have been given and are ineffective, or is no longer eligible for additional standard treatment options.

The study is comprised of a dose escalation phase to determine the maximum tolerated dose and the RP2D and an expansion phase to further explore the safety and preliminary antitumor activity of NB004.

ELIGIBILITY:
Inclusion Criteria:

1. males or females of any race>(=)18 years age.
2. Histologically and/or cytologically confirmed diagnosis of advanced solid tumors that are without standard treatment options (part 1).

   Pathologically confirmed locally advanced or metastatic solid tumors with KRAS G12C mutation as determined by a test that has been approved by FDA or local health authority (part 2&3).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy>(=)12 weeks.
5. Adequate organ and marrow function.
6. Measurable or evaluable disease.

Exclusion Criteria:

1. Prior anti-cancer therapy within 2 weeks or at least 5 half-lives, whichever is longer, up to a maximum of 3 weeks, before the first dose.
2. Toxicities from previous anti-cancer therapy that have not recovered as required.
3. Brain metastatic disease, spinal cord compression, or leptomeningeal carcinomatosis.
4. Active infection including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV):
5. Female subjects who are pregnant, or breastfeeding, or planning to become pregnant while in this study or within 3 months after the last dose.
6. Male subjects who plan to father a child while enrolled in the study or within 3 months after the last dose.
7. Received prior treatment with a PIM kinase inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities----Part 1/2 | When subject complete 1 cycle (28 days) treatment with safety and tolerability assessment by investigators.
  Dose-limiting toxicities will be reviewed as a subset of adverse events that occurs within the first 28 days of dosing and meet protocol-specified criteria.
Incidence of adverse events----Part 1/2 | Approximately 24 months since the first subject enrolled
  An adverse event is any untoward medical occurrence in a participant who received study drug without regard to causal relationship.
Objective Response Rate (ORR) ----Part 3 | [Time Frame: Approximately 24 months since the first subject enrolled]
  Objective Response Rate (ORR) is defined as the percentage of patients whose efficacy is confirmed as complete response (CR) or partial response (PR)
Duration of Response (DOR) ----Part 3 | [Time Frame: Approximately 24 months since the first subject enrolled]
  DOR is defined as the time from the date of first documented response until date of documented progression, for subjects who achieve CR or PR.
Time to Response (TTR) ----Part 3 | [Time Frame: Approximately 24 months since the first subject enrolled]
  TTR is defined as the time interval between the date of first administration and the date of the first recording of response. At the same time, the initial response time and the time to best response will be calculated.
Progression-free Survival (PFS) ----Part 3 | [Time Frame: Approximately 24 months since the first subject enrolled]
  PFS is defined as the time from the date of the first dose until the date of disease progression, as defined by RECIST v1.1, or death.
Clinical Benefit Rate (CBR) ----Part 3 | [Time Frame: Approximately 24 months since the first subject enrolled]
  CBR is defined as the number of subjects with CR or PR or with SD maintained ≥24 weeks (as assessed by the Investigator, using RECIST v1.1) divided by the number of subjects in the analysis. Subjects without a postbaseline tumor assessment will be considered as having no clinical benefit.
Overall survival (OS) ----Part 3 | [Time Frame: Approximately 24 months since the first subject enrolled]
  OS is defined as the time from treatment start with study drug until event of death due to any cause.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax)----Part 1 | Approximately 24 months since the first subject enrolled
  Maximum observed plasma concentration (Cmax)
Time to Cmax (Tmax)----Part 1 | Approximately 24 months since the first subject enrolled
  Time to Cmax (Tmax)
Area under the curve (AUC) from time zero to the last measurable concentration AUC (0-t) ----Part 1 | Approximately 24 months since the first subject enrolled
  AUC (0-t) = Area under the serum concentration versus time curve from time zero (pre-dose) to the time of the last
Terminal elimination half life----Part 1 | Approximately 24 months since the first subject enrolled
  Terminal elimination half life
Objective Response Rate (ORR)----Part 2 | Approximately 24 months since the first subject enrolled
  Objective Response Rate (ORR) is defined as the percentage of patients whose efficacy is confirmed as complete response(CR) or partial responses(PR)
Duration of Response(DOR)----Part 2 | Approximately 24 months since the first subject enrolled
  DOR is defined as the time from the date of first documented response until date of documented progression, for subjects who achieve CR or PR.
Clinical Benefit Rate (CBR) ----Part 2 | [Time Frame: Approximately 24 months since the first subject enrolled]
  CBR is defined as the number of subjects with CR or PR or with SD maintained ≥24 weeks (as assessed by the Investigator, using RECIST v1.1) divided by the number of subjects in the analysis. Subjects without a postbaseline tumor assessment will be considered as having no clinical benefit.
Time to Response (TTR) ----Part 2 | [Time Frame: Approximately 24 months since the first subject enrolled]
  TTR is defined as the time interval between the date of first administration and the date of the first recording of response. At the same time, the initial response time and the time to best response will be calculated.
Progression-free Survival (PFS) ----Part 2 | [Time Frame: Approximately 24 months since the first subject enrolled]
  PFS is defined as the time from the date of the first dose until the date of disease progression, as defined by RECIST
Overall survival (OS) ----Part 2 | [Time Frame: Approximately 24 months since the first subject enrolled]
  OS is defined as the time from treatment start with study drug until event of death due to any cause

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - LSU-LCMC Health Cancer Center, New Orleans, Louisiana
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- China (2):
  - National Cheng Kung University Hospital（NCKUH）, Tainan, Taiwan
  - National Taiwan University Hospital Yunlin Branch, Yunlin, Taiwan